CLINICAL TRIAL: NCT02226926
Title: Mechanism of Dipyridamole Action in Platelets: in Vivo Study With Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9.142
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Aspirin, Dipyridamole Drug Combination; Aspirin

ARMS (3):
- Aggrenox (Experimental): Dipyridamole extended release / Acetylsalicylic acid
  Interventions: Drug: Aggrenox
- Persantin Retard (Active Comparator): Dipyridamole extended release
  Interventions: Drug: Persantin Retard
- Acetylsalicylic acid (Active Comparator)
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Aggrenox
  Arms: Aggrenox
Drug: Persantin Retard
  Arms: Persantin Retard
Drug: Acetylsalicylic acid
  Arms: Acetylsalicylic acid

SUMMARY:
Investigation of the mechanism of dipyridamole action in platelets in an in-vivo study with healthy volunteers treated Aggrenox in comparison with volunteers treated with Persantin Retard or Acetylsalicylic Acid using platelet Vasodilator-Stimulated-Phosphoprotein (VASP)-phosphorylation as indication for an action and measurements of dipyridamole plasma levels

ELIGIBILITY:
Inclusion Criteria:

* Healthy females/males
* Age range from 18 to 60
* Volunteers will have given their written informed consent in accordance with local ethics committee and local legislation

Exclusion Criteria:

* Known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the nervous system (such as epilepsy) or with psychiatric disorders or neurological disorders
* Known history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Drug intake with long half-life (> 24 hours), < 1 month prior to administration or during the trial
* Volunteers received any other drugs which might influence the results of the trial, < 10 days prior to administration or during the trial
* Participation in another study with an investigational drug, < 1 month prior to administration or during the trial
* Smoking more than 15 cigarettes or 4 cigars or 4 pipes/day
* Drinking more than 60 g of alcohol per day
* Unable to refrain from excessive consumption of methylxanthine containing drinks or food
* Drug addiction
* Blood donation (> 400 ml), < 4 weeks prior to administration or during the trial
* Participation in excessive physical activities, < 5 days prior to administration or during the trial

For female volunteers:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (acceptable: oral contraceptives, condoms, etc.)
* Lactation period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2000-07; Primary Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
VASP-Ser239 / VASP-Ser157-phosphorylation | up to day 10
  induced by sodium nitroprusside (SNP) 0.5µM or SNP 0.3µM and prostaglandin E1 (PG-E1) 0.3nM (Western Blot)

SECONDARY OUTCOMES:
Change in Dipyridamole plasma levels | up to day 10
  by High Performance Liquid Chromatography (HPLC)